CLINICAL TRIAL: NCT00003380
Title: A Phase I Study of Liposomal Doxorubicin (Doxil) and Prolonged Etoposide As Second Line Therapy in Ovarian, Tubal and Peritoneal Carcinoma
Brief Title: Liposomal Doxorubicin and Etoposide in Treating Patients With Recurrent or Persistent Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066375; GOG-9704
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2002-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Etoposide

INTERVENTIONS:
Drug: etoposide
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy consisting of liposomal doxorubicin and etoposide in treating patients who have recurrent or persistent ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the optimal dose of doxorubicin HCl liposomal and prolonged oral etoposide in patients with recurrent or persistent ovarian, tubal, and peritoneal carcinoma. II. Determine the nature and degree of toxicity of this therapy in these patients. III. Evaluate the response rate of patients with measurable disease.

OUTLINE: This is a dose escalation, multicenter study of etoposide and doxorubicin HCl liposome. Patients receive doxorubicin HCl liposome IV over 1 hour on day 1, followed by oral etoposide for 8-14 days beginning on day 2. For patients who achieve partial or complete response, treatment repeats every 4 weeks for 1 year in the absence of disease progression or unacceptable toxicity. For patients with stable disease, treatment repeats every 4 weeks for 6 months. In the absence of dose limiting toxicity (DLT) in the first 3 patients treated, subsequent cohorts of 3-6 patients each receive doses of etoposide for more prolonged periods. After 14 days of oral etoposide, the dose of doxorubicin HCl liposome is escalated. The maximum tolerated dose is defined as the dose preceding that at which 2 of 6 patients experience DLT. Patients are followed every 3 months for 1 year, then until death.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or persistent ovarian, tubal, or peritoneal carcinoma of the following cell types: Serous adenocarcinoma Mucinous adenocarcinoma Clear cell adenocarcinoma Transitional cell Endometrioid adenocarcinoma Undifferentiated carcinoma Mixed epithelial carcinoma Malignant Brenner tumor Adenocarcinoma not otherwise specified Must not be eligible for any other higher priority phase II or phase III GOG protocol

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT/SGPT/GGT no greater than 2.5 times normal Alkaline phosphatase no greater than 2.5 times normal No acute hepatitis Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance greater than 50 mL/min Cardiovascular: LVEF within normal range as determined by MUGA No congestive heart failure or unstable angina No myocardial infarction within the past 6 months Prior abnormal cardiac conduction (e.g., bundle branch block, heart block) allowed if stable for at least 6 months Other: No significant infection No septicemia Body surface area at least 1 m2 Adequate intestinal function (i.e., does not require IV hydration or nutritional support) No severe gastrointestinal bleeding No other invasive malignancies within the past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy and recovered Chemotherapy: Must have received at least 1 prior cisplatin-paclitaxel based regimen At least 3 weeks since prior chemotherapy and recovered No prior anthracycline therapy Endocrine therapy: At least 3 weeks since prior endocrine therapy and recovered Radiotherapy: No prior radiotherapy to more than 10% of bone marrow Surgery: At least 3 weeks since prior surgery and recovered

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-05; Primary Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — The Cleveland Clinic
Locations (63):
- United States (62):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada